CLINICAL TRIAL: NCT06272877
Title: Effectiveness of Fluidotherapy in Patients With Conservatively Treated Distal Radius Fractures
Brief Title: Fluidotherapy in Patients With Distal Radius Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Levent Horoz, Principal Investigator, Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 129944-54
Record Dates: First submitted 2024-02-16; First posted 2024-02-22 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Distal Radius Fractures; Edema Arm; Pain
Keywords: Distal Radius Fractures; edema; pain; physical therapy; fluidotherapy
MeSH Terms: conditions — Wrist Fractures; Pain; Edema

STUDY DESIGN:
Intervention Model Description: Randomised controlled
Who Masked: Investigator, Outcomes Assessor
Masking Description: The Investigator and the outcomes assesor will be different persons. Statician will be different person.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluidotherapy Group (Experimental): Fluidotherapy will be applied to the group in addition to the conservative rehabilitation program received by the control group. Fluidotherapy will be applied 20 minutes a day, 5 days a week for 4 weeks.
  Interventions: Other: Fluidotherapy; Other: conventional rehabilitation program
- Control group (Active Comparator): Only the conventional rehabilitation program will be applied by a physiotherapist for 6 weeks.
  Interventions: Other: conventional rehabilitation program

INTERVENTIONS:
Other: Fluidotherapy — Fluidotherapy is a dry environment created by mobilizing solid particles using heated air flow. Fluidotherapy will be applied 20 minutes a day, 5 days a week for 4 weeks.
  Arms: Fluidotherapy Group
Other: conventional rehabilitation program — The conventional rehabilitation program determined before the study will be implemented by a physiotherapist in the hospital for 6 weeks.

SUMMARY:
Distal radius fractures are the most common fractures when looking at upper extremity fractures. The incidence of distal radius fractures is increasing day by day, and when looking at the databases of various countries, its annual prevalence reaches 70,000 in the UK and 640,000 in the USA. Most of these fractures are related to osteoporosis and require appropriate treatment. If not, it causes loss of work force, permanent disability, and limitation in daily activities.

Fluidotherapy has also proven to be effective in reducing hand edema in patients with carpal tunnel syndrome and stroke, examining its effect on nerve conduction velocities, and warming hypothermic patients. Compared to these treatment methods, fluid therapy reduces both joint capsule and muscle temperature by 9°C and 5.7°C, respectively. has been reported to increase.

DETAILED DESCRIPTION:
Reducing pain and edema after Distal Radius fracture is an important part of postoperative rehabilitation. Various massage and mobilization methods were applied to this patient population in the postoperative period. In a recent study evaluating the effectiveness of Whirlpool treatment, it was reported that studies on the effectiveness of fluidotherapy are also needed. There is no study in the literature evaluating the effectiveness of fluidotherapy in the postoperative rehabilitation program in patients who underwent surgery for distal radius fractures.

This study aimed to evaluate the effect of adding fluidotherapy to the early rehabilitation program on pain, edema, joint range of motion and functionality after the cast is removed in patients who received conservative cast treatment due to distal radius fracture.

ELIGIBILITY:
Inclusion Criteria:

-Treating with a cast due to distal radius fracture being over 18 years old

Exclusion Criteria:

* Presence of polytrauma
* History of previous limb-related surgery
* Hemiplegia in the involved limb
* Contracture in the involved limb
* Arterial and venous occlusions
* Lymphatic system disorders
* Heart and circulatory system disorders
* Hepatitis, Measles, Sepsis infectious diseases or fever
* Open wound on the applied hand.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | Baseline
  Visual analog scale (VAS) was used for pain assessment. VAS is a 10-point Likert scale.A score of 0 indicates the best result, a score of 10 indicates the worst result. Higher scores indicate higher pain.
Visual analog scale | 2th week
  Visual analog scale (VAS) was used for pain assessment. VAS is a 10-point Likert scale.A score of 0 indicates the best result, a score of 10 indicates the worst result. Higher scores indicate higher pain.
Visual analog scale | 6th week
  Visual analog scale (VAS) was used for pain assessment. VAS is a 10-point Likert scale.A score of 0 indicates the best result, a score of 10 indicates the worst result. Higher scores indicate higher pain.
Wrist joint range of motion | Baseline
  Wrist joint range of motion: Measurement of wrist joint range of motion (ROM) with a goniometer is the most frequently used method in clinical practice that provides objective evaluation and error-free measurement. In our study, wrist ROM measurements will be made with a goniometer using the neutral zero method. This method is a painless and non-invasive measurement method.
Wrist joint range of motion | 2th week
  Wrist joint range of motion: Measurement of wrist joint range of motion (ROM) with a goniometer is the most frequently used method in clinical practice that provides objective evaluation and error-free measurement. In our study, wrist ROM measurements will be made with a goniometer using the neutral zero method. This method is a painless and non-invasive measurement method.
Wrist joint range of motion | 6th week
  Wrist joint range of motion: Measurement of wrist joint range of motion (ROM) with a goniometer is the most frequently used method in clinical practice that provides objective evaluation and error-free measurement. In our study, wrist ROM measurements will be made with a goniometer using the neutral zero method. This method is a painless and non-invasive measurement method.
Circumference (mm) | Baseline
  Environmental Measurement; the both hands and wrists of the patient will be measured with the help of a tape measure using the figure of eight method. The cm difference between both upper extremities will be recorded.
Circumference (mm) | 2th week
  Environmental Measurement; the both hands and wrists of the patient will be measured with the help of a tape measure using the figure of eight method. The cm difference between both upper extremities will be recorded.
Circumference (mm) | 6th week
  Environmental Measurement; the both hands and wrists of the patient will be measured with the help of a tape measure using the figure of eight method. The cm difference between both upper extremities will be recorded.

SECONDARY OUTCOMES:
Gross Grip Strength: | Baseline
  Jamar dynamometer wii use to evaluate gross grip strength.Higher values indicate increased grip strength
Gross Grip Strength: | 2th week
  Jamar dynamometer wii use to evaluate gross grip strength.Higher values indicate increased grip strength
Gross Grip Strength: | 6th week
  Jamar dynamometer wii use to evaluate gross grip strength.Higher values indicate increased grip strength
Patient-Rated Wrist Evaluation (PRWE) questionnaire | Baseline
  Patient-Rated Wrist Evaluation (PRWE) questionnaire: PRWE is a 15-item questionnaire.High scores indicate functional impairment designed to measure wrist pain and disability in activities of daily living.The maximum score that can be obtained from the pain subscale is 50 and the minimum is 0.
  The maximum score that can be obtained from the function subscale is 50 and the minimum is 0.
Patient-Rated Wrist Evaluation (PRWE) questionnaire | 2th week
  Patient-Rated Wrist Evaluation (PRWE) questionnaire: PRWE is a 15-item questionnaire.High scores indicate functional impairment designed to measure wrist pain and disability in activities of daily living.The maximum score that can be obtained from the pain subscale is 50 and the minimum is 0.
  The maximum score that can be obtained from the function subscale is 50 and the minimum is 0.
Patient-Rated Wrist Evaluation (PRWE) questionnaire | 6th week
  Patient-Rated Wrist Evaluation (PRWE) questionnaire: PRWE is a 15-item questionnaire.High scores indicate functional impairment designed to measure wrist pain and disability in activities of daily living.The maximum score that can be obtained from the pain subscale is 50 and the minimum is 0.
  The maximum score that can be obtained from the function subscale is 50 and the minimum is 0.

CONTACTS AND LOCATIONS:
Overall Officials: Levent Horoz, Asst Prof, Principal Investigator — Kirsehir Research and Training Hospital
Locations (1):
- Kirsehir Research and Training Hospital, Kırşehir, Kişrsehşr, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szekeres M, MacDermid JC, Grewal R, Birmingham T. The short-term effects of hot packs vs therapeutic whirlpool on active wrist range of motion for patients with distal radius fracture: A randomized controlled trial. J Hand Ther. 2018 Jul-Sep;31(3):276-281. doi: 10.1016/j.jht.2017.08.003. Epub 2017 Oct 12. PMID 28893496
- [Background] Gutierrez-Espinoza H, Araya-Quintanilla F, Olguin-Huerta C, Valenzuela-Fuenzalida J, Gutierrez-Monclus R, Moncada-Ramirez V. Effectiveness of manual therapy in patients with distal radius fracture: a systematic review and meta-analysis. J Man Manip Ther. 2022 Feb;30(1):33-45. doi: 10.1080/10669817.2021.1992090. Epub 2021 Oct 20. PMID 34668847
- [Background] Borrell RM, Parker R, Henley EJ, Masley D, Repinecz M. Comparison of in vivo temperatures produced by hydrotherapy, paraffin wax treatment, and Fluidotherapy. Phys Ther. 1980 Oct;60(10):1273-6. doi: 10.1093/ptj/60.10.1273. PMID 7443789